CLINICAL TRIAL: NCT04738110
Title: Post-operative Imaging in High Grade Glioma: is Management Influenced?
Acronym: PIGMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH20-139
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KCH patients: 75 high grade glioma patients from KCH
  Interventions: Other: MRI
- NHNN patients: 75 high grade glioma patients from NHNN
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Structural MR (T2, FLAIR, T1 and T1+C), DCE, DSC

SUMMARY:
Magnetic resonance imaging (MRI) is likely to play an important role in the management of high grade glioma. Appropriate and timely neuroimaging in the follow up period is believed to be crucial in making subsequent management decisions. However, there is a paucity in the literature providing evidence to support this. The aim of this study is to determine whether neuroimaging performed at each component of the patient pathway after initial high grade glioma treatment, actually results in a real change in management (as opposed to a perceived change in management). The main emphasis is on all imaging used at the time of a MDM, however, we will also study specifically dynamic susceptibility contrast-enhanced (DSC) MRI and dynamic contrast enhanced (DCE) MRI.

The study is in the format of Mock MDMs to be compatible with real life decision making. Using retrospective identical information available at the MDM i.e. compiled recent correspondence, histopathological and molecular information, the MDM members (oncology nurse, oncologist, neurosurgeon, neuroradiologist, pathologist/molecular scientist) will prospectively determine the patient management with and without the imaging.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven HGG patients (Grade III and IV WHO criteria)
* Underwent surgery, radiotherapy and chemotherapy regimen according to 2018 NICE guidelines (1)
* >=18 years old
* Has follow-up MRI imaging (T1, T2, FLAIR and T1 with contrast enhancement) and also DSC and DCE imaging
* Evaluated at MDT meetings between March 2018 and March 2020.

Exclusion Criteria:

* Patients who have insufficient clinical and radiological follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HGG (Grade III and IV WHO criteria) patients discussed in MDTM between March 2018 and March 2020 at KCH and NHNN are being studied.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-12-16 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Determine how MR imaging influences the management of HGG patients | 12 months

SECONDARY OUTCOMES:
Determine how advanced MR imaging influences the management of HGG patients | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- King´s College Hospital NHS Foundation trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No